CLINICAL TRIAL: NCT01518244
Title: Assessing the Efficacy and Tolerability of AZARGA® (Brinzolamide 1%/Timolol 0.5% Fixed Combination) as Replacement Therapy in Patients on Brimonidine 0.2%/Timolol 0.5% Fixed Combination Therapy (COMBIGAN®) in Latin America
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RDG-11-198
Record Dates: First submitted 2012-01-23; First posted 2012-01-25 (Estimated); Results first posted 2014-04-04 (Estimated); Last update posted 2015-08-07 (Estimated); Status verified 2014-02

CONDITIONS: Glaucoma
Keywords: Primary open angle-glaucoma; Ocular hypertension; Pigment dispersion glaucoma
MeSH Terms: conditions — Glaucoma; Glaucoma, Open-Angle; Ocular Hypertension | interventions — brinzolamide; Azarga

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- AZARGA® (Experimental): Brinzolamide/timolol maleate fixed combination, 1 drop self-administered in study eye(s) twice a day for 8 weeks
  Interventions: Drug: Brinzolamide/timolol maleate fixed combination

INTERVENTIONS:
Drug: Brinzolamide/timolol maleate fixed combination
  Other Names: AZARGA®

SUMMARY:
The purpose of this study was to assess the efficacy and tolerability of changing to AZARGA® from prior COMBIGAN® pharmacotherapy in participants with open-angle glaucoma or ocular hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of ocular hypertension, exfoliative open-angle glaucoma, or pigment dispersion glaucoma in at least one eye (study eye).
* On a stable IOP (intra-ocular pressure) lowering regimen within 30 days of Screening Visit.
* IOP considered safe in both eyes in order to assure clinical stability of vision and optic nerve throughout the study period.
* Best corrected visual acuity of 6/60 (20/200 Snellen; 1.0 LogMAR) or better in each eye.
* IOP between 19 and 35 mmHG in at least one eye (which would be the study eye) while on brimonidine/timolol fixed combination therapy.
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Presence of other primary or secondary glaucoma.
* History of ocular herpes simplex.
* Any abnormality preventing reliable applanation tonometry.
* Corneal dystrophies.
* Concurrent infectious/noninfectious conjunctivitis, keratitis, or uveitis in either eye. Blepharitis or non-clinically significant conjunctival injection is allowed.
* Intraocular conventional surgery or laser surgery in study eye(s) less than three months prior to Screening Visit.
* Risk of visual field or visual acuity worsening as a consequence of participation in the study, in the opinion of the investigator.
* Progressive retinal or optic nerve disease from any cause.
* Use of systemic medications known to affect IOP which have not been on a stable course for 7 days prior to Screening Visit or an anticipated change in the dosage during the course of the study.
* Pregnant or lactating.
* Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2011-12; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Doug Hubatsch, Study Director — Alcon Research

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 6 study centers located in South America: Argentina (3), Chile (1), and Mexico (2).
Pre-assignment Details: This reporting group includes all participants who received at least one dose of AZARGA®.
Period: Overall Study
Arm/Group | AZARGA®
Started | 50
Completed | 47
Not Completed | 3
Not completed — Adverse Event | 3

BASELINE CHARACTERISTICS:
Population: The analysis population includes all participants who received AZARGA® and with at least one on-therapy study visit (V2 or V3). Of the 50 enrolled, 1 participant discontinued after V1 and before V2.
Arm/Group | AZARGA®
Number analyzed (Participants) | 49
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.67 (11.51)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30
  Male | 19

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Intraocular Pressure (IOP) From Baseline (Prior Therapy) at Week 8
Description: IOP (fluid pressure inside the eye) was measured by Goldmann applanation tonometry. A higher IOP can be a greater risk for developing glaucoma or glaucoma progression (leading to optic nerve damage). A more negative change indicates a greater amount of improvement. One eye was chosen as the study eye, and only data from the study eye were used for the efficacy analysis.
Time Frame: Baseline, Week 8
Population: The analysis population includes all participants who received AZARGA® and with at least 1 on-therapy study visit (V2 or V3).
Measure: Mean (Standard Deviation); unit: milllimeters mercury (mmHg)
Arm/Group | AZARGA®
Number analyzed (Participants) | 49
milllimeters mercury (mmHg) | -3.60 (3.01)

2. Secondary Outcome: Percentage of Subjects Who Reach Target IOP (≤18 mmHg) at Week 8
Description: IOP (fluid pressure inside the eye) was measured by Goldmann applanation tonometry. A higher IOP can be a greater risk for developing glaucoma or glaucoma progression (leading to optic nerve damage). One eye was chosen as the study eye, and only data from the study eye were used for the efficacy analysis.
Time Frame: Week 8
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | AZARGA®
Number analyzed (Participants) | 49
percentage of participants | 55.3

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected for the duration of the study (December 2011-February 2013). An AE was defined as any untoward medical occurrence in a subject administered the test product, regardless of causal relationship with such product.
Description: The analysis population includes all participants who received at least one dose of AZARGA®.
Arm/Group | AZARGA®
Serious Adverse Events (participants affected / at risk) | 0/50
Other Adverse Events (participants affected / at risk) | 4/50
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AZARGA® (N=50)
Eye irritation (Eye disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.